CLINICAL TRIAL: NCT00183274
Title: Short-term Versus Long-term Treatment in Generalized Anxiety Disorder
Brief Title: Effectiveness of Long-Term Versus Short-Term Treatment of Generalized Anxiety Disorder With Venlafaxine XR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Karl Rickels, Professor of Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MH65963; R01MH065963 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Anxiety Disorders
Keywords: Generalized Anxiety Disorder; Chronic Mediation Treatment; Double-Blind; Placebo Controlled; Venlafaxine XR; Relapse
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Recurrence | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Open-Label Group (Active Comparator): 6-month randomized phase of Venlafaxine XR at a flexible dose of 75 - 225 mg/d
  Interventions: Drug: Venlafaxine XR
- Double-Blind Drug Group (Active Comparator): 6-month randomized, double-blind phase of Venlafaxine XR at a flexible dose of 75 - 225 mg/d occurring between months 6 - 12 of the study
  Interventions: Drug: Venlafaxine XR
- Double-Blind Placebo Group (Placebo Comparator): 6-month randomized, double blind phase of placebo occurring between months 6 - 12 of the study
  Interventions: Drug: Placebo
- Double-Blind Drug-After-Drug Group (Active Comparator): 6-month randomized, double blind phase of Venlafaxine XR at a flexible dose of 75 - 225 mg/d occurring between months 13 - 19 of the study
  Interventions: Drug: Venlafaxine XR
- Double-Blind Placebo-After-Drug Group (Placebo Comparator): 6-month randomized, double blind phase of placebo occurring between months 13 - 19 of the study
  Interventions: Drug: Placebo
- Double-Blind Placebo-After-Placebo Group (Placebo Comparator): 6-month randomized, double blind phase of placebo occurring between months 13 - 19 of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Venlafaxine XR — Six month intervention of Venlafaxine XR treatment with flexible range of 75 to 225 mg/d
  Other Names: selective serotonin and norepinephrine reuptake inhibitors; Effexor; Effexor XR; Venlafaxine hydrochloride extended release; Trevilor; Lanvexin
  Arms: Double-Blind Drug Group; Double-Blind Drug-After-Drug Group; Open-Label Group
Drug: Placebo — six month intervention with placebo drug
  Arms: Double-Blind Placebo Group; Double-Blind Placebo-After-Drug Group; Double-Blind Placebo-After-Placebo Group

SUMMARY:
This study will assess the effectiveness of venlafaxine XR, randomized to either venlafaxine XR or placebo in preventing the relapse of generalized anxiety disorder after 6 months of treatment versus 12 months of treatment.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is a highly prevalent, chronic psychiatric disorder. Despite the fact that GAD frequently demands prolonged treatment with medication, very little is known about the benefits of long-term treatment. GAD is characterized by 6 months or more of exaggerated worry and tension that is unfounded or much more severe than the normal anxiety most people experience. People with GAD are unable to relax and often suffer from insomnia. Venlafaxine XR, a drug used to treat depression, has been shown to be effective in the short-term treatment of GAD. However, its benefits over a course of more than 8 weeks have not been assessed. This study will evaluate the effectiveness of venlafaxine XR in treating GAD on a long-term basis and preventing the relapse of GAD after 6 months of treatment versus 12 months of treatment.

Participants in this double-blind study will first receive 6 months of open-label treatment with venlafaxine XR. Upon completion of this initial phase, participants will be randomly assigned to either continue on venlafaxine XR or begin taking placebo. After 12 months, participants taking venlafaxine XR will be randomly assigned to continue on the drug or switch to placebo. Participants will have 22 study visits over at least 18 months. Follow-up visits will occur 24 months after enrollment. Relapse of GAD will be assessed with the Hamilton Anxiety Scale and Global Severity and Improvement Scale. A variety of methods, including questionnaires and standardized scales, will be used to assess secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* GAD diagnosis by structured interview
* Hamilton Anxiety Scale score of 18 or MORE
* Clinical Global Impressions Severity Scale score of at least 4
* Hamilton Depression Scale score of 18 or less
* Hamilton Depression Scale suicide item score less than 2
* Use of an effective form of contraception throughout the study

Exclusion Criteria:

* Hypersensitivity to venlafaxine XR
* History of seizures
* Episode of major depressive disorder in the previous 6 months
* History of any psychotic illness, bipolar disorder, or dementia
* Substance abuse and dependence during the past 6 months
* Other anxiety disorders with the exception of social phobia as long as GAD is primary
* Regular use of anxiolytics or antidepressants within 7 days of study onset
* Use of fluoxetine or monoamine oxidase inhibitors within 28 days of study onset (low dose usage of benzodiazepines will not prevent participation)
* Use of other psychotropic medication besides benzodiazepines during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2004-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Rickels, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, 3535 Market Street, Suite 670, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rickels K, Etemad B, Rynn MA, Lohoff FW, Mandos LA, Gallop R. Remission of generalized anxiety disorder after 6 months of open-label treatment with venlafaxine XR. Psychother Psychosom. 2013;82(6):363-71. doi: 10.1159/000351410. Epub 2013 Sep 20. PMID 24061331
- [Result] Rickels K, Etemad B, Khalid-Khan S, Lohoff FW, Rynn MA, Gallop RJ. Time to relapse after 6 and 12 months' treatment of generalized anxiety disorder with venlafaxine extended release. Arch Gen Psychiatry. 2010 Dec;67(12):1274-81. doi: 10.1001/archgenpsychiatry.2010.170. PMID 21135327
- [Derived] Jung J, Tawa EA, Muench C, Rosen AD, Rickels K, Lohoff FW. Genome-wide association study of treatment response to venlafaxine XR in generalized anxiety disorder. Psychiatry Res. 2017 Aug;254:8-11. doi: 10.1016/j.psychres.2017.04.025. Epub 2017 Apr 14. PMID 28437668
- [Derived] Saung WT, Narasimhan S, Lohoff FW. Lack of influence of DAT1 and DRD2 gene variants on antidepressant response in generalized anxiety disorder. Hum Psychopharmacol. 2014 Jul;29(4):316-21. doi: 10.1002/hup.2404. Epub 2014 Apr 10. PMID 24723432
- [Derived] Cooper AJ, Narasimhan S, Rickels K, Lohoff FW. Genetic polymorphisms in the PACAP and PAC1 receptor genes and treatment response to venlafaxine XR in generalized anxiety disorder. Psychiatry Res. 2013 Dec 30;210(3):1299-300. doi: 10.1016/j.psychres.2013.07.038. Epub 2013 Aug 22. PMID 23972788
- [Derived] Cooper AJ, Rickels K, Lohoff FW. Association analysis between the A118G polymorphism in the OPRM1 gene and treatment response to venlafaxine XR in generalized anxiety disorder. Hum Psychopharmacol. 2013 May;28(3):258-62. doi: 10.1002/hup.2317. Epub 2013 May 8. PMID 23658070
- [Derived] Lohoff FW, Narasimhan S, Rickels K. Interaction between polymorphisms in serotonin transporter (SLC6A4) and serotonin receptor 2A (HTR2A) genes predict treatment response to venlafaxine XR in generalized anxiety disorder. Pharmacogenomics J. 2013 Oct;13(5):464-9. doi: 10.1038/tpj.2012.33. Epub 2012 Aug 21. PMID 22907732
- [Derived] Narasimhan S, Aquino TD, Multani PK, Rickels K, Lohoff FW. Variation in the catechol-O-methyltransferase (COMT) gene and treatment response to venlafaxine XR in generalized anxiety disorder. Psychiatry Res. 2012 Jun 30;198(1):112-5. doi: 10.1016/j.psychres.2011.12.034. Epub 2012 Mar 13. PMID 22417933
- [Derived] Lohoff FW, Aquino TD, Narasimhan S, Multani PK, Etemad B, Rickels K. Serotonin receptor 2A (HTR2A) gene polymorphism predicts treatment response to venlafaxine XR in generalized anxiety disorder. Pharmacogenomics J. 2013 Feb;13(1):21-6. doi: 10.1038/tpj.2011.47. Epub 2011 Oct 18. PMID 22006095
- [Derived] Narasimhan S, Aquino TD, Hodge R, Rickels K, Lohoff FW. Association analysis between the Val66Met polymorphism in the brain-derived neurotrophic factor (BDNF) gene and treatment response to venlafaxine XR in generalized anxiety disorder. Neurosci Lett. 2011 Oct 10;503(3):200-2. doi: 10.1016/j.neulet.2011.08.035. Epub 2011 Aug 26. PMID 21889574

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Most patients (n=239) were recruited and seen by Penn research psychiatrists in 4 primary care practices; others (n=95) responded to media advertising (radio & print ads) at the central clinic at the University of Pennsylvania
Pre-assignment Details: 7-day washout period of any psychoactive medication;other antidepressants and herbal products. Subject on certain medications, such as monamine oxidase inhibitor, investigational and antipsychotic drugs had to be off these medications for at least 30 days.
Groups:
- Phase 1: Open-Label: Patients received 75mg - 225 mg of open-label venlafaxine XR for 6 months.
- Phase 2: Double-Blind Venlafaxine XR: Responders to 6 months of open-label venlafaxine XR treatment were randomized to double-blind treatment in 60:40 ratio of drug to placebo
- Phase 2: Double-Blind Placebo: Responders to 6 months of open-label venlafaxine XR treatment were randomized to double-blind treatment in a 60:40 ratio of drug to placebo
- Phase 3: Double-Blind Relapse Phase (Drug After Drug): Patients administered venlafaxine XR in phase 2 continued to take the drug during phase 3
- Phase 3: Double-Blind Relapse Phase (Placebo After Drug): Patients administered venlafaxine XR in Phase 2 were given a placebo in Phase 3
- Phase 3: Double-Blind Relapse Phase (Placebo After Placebo): Patients administered placebo in Phase 2 continued to take placebo during Phase 3
Period: Phase 1: Open-Label
Arm/Group | Phase 1: Open-Label | Phase 2: Double-Blind Venlafaxine XR | Phase 2: Double-Blind Placebo | Phase 3: Double-Blind Relapse Phase (Drug After Drug) | Phase 3: Double-Blind Relapse Phase (Placebo After Drug) | Phase 3: Double-Blind Relapse Phase (Placebo After Placebo)
Started | 268 | 0 | 0 | 0 | 0 | 0
Completed | 158 (110 dropouts during phase 1) | 0 | 0 | 0 | 0 | 0
Not Completed | 110 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 31 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 13 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 11 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 33 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 9 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: Double-Blind
Arm/Group | Phase 1: Open-Label | Phase 2: Double-Blind Venlafaxine XR | Phase 2: Double-Blind Placebo | Phase 3: Double-Blind Relapse Phase (Drug After Drug) | Phase 3: Double-Blind Relapse Phase (Placebo After Drug) | Phase 3: Double-Blind Relapse Phase (Placebo After Placebo)
Started | 0 (This phase ended after 6 months. There were no longer participants in this phase.) | 82 (22 did not enter phase 2 due to lack of efficacy and withdrawal of consent) | 54 (22 did not enter phase 2 due to lack of efficacy and withdrawal of consent) | 0 | 0 | 0
Completed | 0 | 56 (8 lost to relapse, 18 lost to dropout) | 11 (29 lost to relapse, 14 lost to dropout) | 0 | 0 | 0
Not Completed | 0 | 26 | 43 | 0 | 0 | 0
Not completed — Relapsed | 0 | 8 | 29 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 18 | 14 | 0 | 0 | 0
Period: Phase 3: Double-Blind
Arm/Group | Phase 1: Open-Label | Phase 2: Double-Blind Venlafaxine XR | Phase 2: Double-Blind Placebo | Phase 3: Double-Blind Relapse Phase (Drug After Drug) | Phase 3: Double-Blind Relapse Phase (Placebo After Drug) | Phase 3: Double-Blind Relapse Phase (Placebo After Placebo)
Started | 0 | 0 (Phase 2 ended at the end of 12 months of study.) | 0 (Phase 2 ended at the end of 12 months of study.) | 15 (8 completed Phase 2 but did not enter phase 3) | 34 (8 completed Phase 2 but did not enter phase 3) | 10 (8 completed Phase 2 but did not enter phase 3)
Completed | 0 | 0 | 0 | 13 (1 lost to relapse and 1 lost to dropout) | 14 (11 lost to relapse and 9 lost to dropout) | 6 (2 lost to relapse and 2 lost to dropout)
Not Completed | 0 | 0 | 0 | 2 | 20 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 9 | 2
Not completed — Relapsed | 0 | 0 | 0 | 1 | 11 | 2

BASELINE CHARACTERISTICS:
Population: 334 participants were consented, but 64 withdrew consent and 2 deviated from protocol, resulting in 268 participants who entered the initial Phase 1.
Groups:
- Venlafaxine XR: Venlafaxine XR flexible dose of 75 - 225 mg/d
  Venlafaxine XR : All participants will take venlafaxine for 6 months. After this initial 6 months, participants who are not randomized to placebo will continue to take venlafaxine.
Arm/Group | Venlafaxine XR
Number analyzed (Participants) | 334
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 280
  >=65 years | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.11 (16.14)
Gender [Count of Participants; unit: Participants]
  Female | 210
  Male | 124
Region of Enrollment [Number; unit: participants]
  United States | 334

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Anxiety
Description: Hamilton Rating Scale for Anxiety - The assessment of anxiety states by rating
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Time Frame: Measured at Months 6 (Open Label), 12 (Double-Blind), and 18 (Double-Blind Relapse)
Population: The primary efficacy analytic method was time-to-relapse analyses estimated using a discrete-time Cox proportional hazards model.
Measure: Mean (Standard Deviation); unit: HAM-A Rating Score
Groups:
- Open-Label: Venlafaxine XR: A 6-month open label administration of flexible dose Venlafaxine XR that occurred between months 1 - 6 of study.
- Double-Blind Venlafaxine XR: A 6-month double-blind administration of Venlafaxine XR that occurred between months 7 - 12.
- Double-Blind Placebo: A 6-month double-blind administration of placebo that occurred between months 7 - 12.
- Double-Blind Relapse Drug After Drug: A 6-month double-blind administration of Venlafaxine XR that occurred between months 13 - 18.
- Double-Blind Relapse Placebo After Drug; Double-Blind Placebo After Placebo: A 6-month double-blind administration of placebo that occurred between months 13 - 18.
Arm/Group | Open-Label: Venlafaxine XR | Double-Blind Venlafaxine XR | Double-Blind Placebo | Double-Blind Relapse Drug After Drug | Double-Blind Relapse Placebo After Drug | Double-Blind Placebo After Placebo
Number analyzed (Participants) | 268 | 82 | 54 | 15 | 34 | 10
HAM-A Rating Score | 4.17 (3.10) | 6.29 (5.44) | 11.35 (5.51) | 5.80 (4.95) | 8.42 (6.12) | 6.19 (5.76)

2. Secondary Outcome: Clinical Global Impressions, Severity of Illness
Description: The CGI provides an overall clinician-determined summary measure that takes into account a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.
  The CGI is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  Results of the "Placebo After Placebo" group in Phase 3 were not entered due to sample size limitations.
Time Frame: Measured at Months 6 (Open Label), 12 (Double-Blind), 18 (Double-Blind, and 24 (Double-Blind Relapse)
Population: The primary efficacy analytic method was time to relapse analyses estimated using a discrete time Cox proportional hazards model.Chisquare analyses were used to contrast relapse or responder rates. In the case of small cell sizes, Fisher exact test replaced chisquare analysis.
Measure: Mean (Standard Deviation); unit: Severity Score
Groups:
- Phase 1: Open-Label Venlafaxine XR: A 6-month administration of Venlafaxine XR that occurred between months 1 - 6 of study.
- Phase 2: Double-Blind Venlafaxine XR: after receiving drug in phase 1, patients continued to receive drug in phase 2
- Phase 2: Double-Blind Placebo: After receiving drug in Phase 1, patients began receiving placebo in phase 2
- Phase 3: Double-Blind Drug After Drug: after receiving drug in phases 1 and 2, patients continued to receive drug in phase 3
- Phase 3: Placebo After Drug: after receiving drug in phases 1 and 2, patients received placebo in phase 3
- Placebo After Placebo: after receiving drug in phases 1 and placebo in phase 2, patients received placebo in phase 3
Arm/Group | Phase 1: Open-Label Venlafaxine XR | Phase 2: Double-Blind Venlafaxine XR | Phase 2: Double-Blind Placebo | Phase 3: Double-Blind Drug After Drug | Phase 3: Placebo After Drug | Placebo After Placebo
Number analyzed (Participants) | 268 | 82 | 54 | 15 | 34 | 10
Severity Score | 1.37 (0.65) | 1.73 (1.27) | 2.64 (1.25) | 1.86 (1.01) | 2.25 (1.17) | 1.95 (1.31)

ADVERSE EVENTS:
Groups:
- Venlafaxine XR: Adverse events were expected with venlafaxine XR. AEs were reported at least once by at least 5% of the study population for all patients who entered treatment. None of the adverse events that were expected or that occurred were considered serious or life threatening.
Arm/Group | Venlafaxine XR
Serious Adverse Events (participants affected / at risk) | 0/268
Other Adverse Events (participants affected / at risk) | 219/268
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Venlafaxine XR (N=268)
Abdominal Pain (General disorders) | 26
Constipation (Gastrointestinal disorders) | 77
Decreased Orgasm (General disorders) | 55
Decreased Sex Drive (General disorders) | 68
Delayed Orgasm (General disorders) | 19
Diarrhea (Gastrointestinal disorders) | 35
Drowsiness (General disorders) | 111
Dry mouth (General disorders) | 130
Faintness (General disorders) | 21
Fatigue (General disorders) | 76
Flatulence (Gastrointestinal disorders) | 66
Gas (Gastrointestinal disorders) | 18
Headache (General disorders) | 97
Increased sweating (General disorders) | 91
Insomnia (General disorders) | 82
Jitteriness (General disorders) | 74
Lightheadedness (General disorders) | 104
Muscle Aches (General disorders) | 50
Nausea (General disorders) | 89
Nightmares (General disorders) | 78

LIMITATIONS AND CAVEATS:
Increased attrition occurring as a function of trial length

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No